CLINICAL TRIAL: NCT00751192
Title: Effect of an Online Video-Based Intervention to Increase HIV Testing in Men Who Have Sex With Men in Peru
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NGO Via Libre (Other)
Collaborators: University of Washington (Other)
Responsible Party: Dr. Magaly Blas, NGO Via Libre and University of Washington
Allocation: Randomized | Model: Single Group | Purpose: Screening
Other Study IDs: 07-6194-J
Record Dates: First submitted 2008-09-10; First posted 2008-09-11 (Estimated); Last update posted 2008-10-09 (Estimated); Status verified 2008-09

CONDITIONS: HIV Infections
Keywords: Men who have sex with men; Peru; HIV testing; video; online; Internet; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Homosexuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Device: HIV-testing motivational videos
- B (Active Comparator)
  Interventions: Device: Standard public health text

INTERVENTIONS:
Device: HIV-testing motivational videos
  Arms: A
Device: Standard public health text
  Arms: B

SUMMARY:
Men who have sex with men (MSM) account for the greatest burden of the HIV and Sexually Transmitted Infection (STI) epidemic in Peru. Current interventions that promote early identification and treatment of these diseases target a limited number of this population because they rely solely on peer education. To assess the use of the Internet as an alternative tool to reach this population the investigators propose to conduct an online randomized controlled trial to compare the effect of HIV-testing motivational videos versus standard public health text, both offered through gay websites. The methodology the investigators will use is divided in: (1) the development period, where the investigators will select gay websites for banner advertisement, create and refine effective recruitment messages and design the online survey and the video-based intervention (2) the intervention period, where participants who meet the eligibility criteria will be randomized into a video or a standard public health text. The videos will be customized for three audiences based on self-identification: gay, non-gay and trans and will be framed within the health-belief model and the stages of change theory (3) in the outcome evaluation period we will compare the 'intentions to get tested' and 'time to HIV testing at the clinic' among MSM of each of the trial arms. If the Internet is an effective venue to reach MSM for HIV testing, Peruvian health programs that target this population may start considering the delivery of web-based interventions and other online prevention services to this under served and hard-to-reach population.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older
* Be a man and report having had sex with a man
* Be a resident of Lima, Peru
* Answer the survey from Lima, Peru
* Have not been tested for HIV during the last year
* Have an email address that when typed twice matched and
* Do not report being HIV positive

Exclusion Criteria:

* Do not meet the inclusion criteria specified above

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2007-10; Primary Completion 2008-04 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Time to HIV testing at the clinic

SECONDARY OUTCOMES:
Intentions to get tested for HIV

CONTACTS AND LOCATIONS:
Locations (1):
- NGO Via Libre, Lima, Lima Province, Peru

REFERENCES:
- [Background] Blas MM, Alva IE, Cabello R, Garcia PJ, Carcamo C, Redmon M, Kimball AM, Ryan R, Kurth AE. Internet as a tool to access high-risk men who have sex with men from a resource-constrained setting: a study from Peru. Sex Transm Infect. 2007 Dec;83(7):567-70. doi: 10.1136/sti.2007.027276. Epub 2007 Oct 11. PMID 17932128
- [Derived] Blas MM, Alva IE, Carcamo CP, Cabello R, Goodreau SM, Kimball AM, Kurth AE. Effect of an online video-based intervention to increase HIV testing in men who have sex with men in Peru. PLoS One. 2010 May 3;5(5):e10448. doi: 10.1371/journal.pone.0010448. PMID 20454667